CLINICAL TRIAL: NCT01891149
Title: Ultrasonographic and Hormonal Characteristics of Malawian Women With and Without Obstetric Fistula
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Jennifer Tang, MD, MSCR, Research Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 12-1880
Record Dates: First submitted 2013-06-25; First posted 2013-07-02 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Obstetric Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Malawian women: Malawian women who present for care at the Fistula Care Centre

SUMMARY:
This study is a cross-sectional study of 110 Malawian women to compare the ultrasonographic and hormonal characteristics of women and without obstetric fistula.

Hypothesis #1: Women with obstetric fistula have a mean cervical length measurement that is at least 10 mm shorter than the mean cervical length measurement of similar women without obstetric fistula.

Hypothesis #2: Evaluation of the hormonal and ultrasonographic characteristics of women with obstetric fistula will allow us to assess the cause of amenorrhea in these women.

DETAILED DESCRIPTION:
This study is a cross-sectional study of 110 Malawian women who present for medical evaluation at the Fistula Care Centre in Lilongwe, Malawi. If a woman enrolls in the study, her demographic, medical history, physical exam, and lab data will be abstracted from her medical records at the Fistula Centre. She will also a pelvic ultrasound on each participant so that the characteristics of her cervix, uterus, and ovaries (such as the cervical length, endometrial thickness and ovarian volume) can be evaluated. If the participant has an obstetric fistula, she will also complete an additional blood draw for lab testing. The laboratory tests will evaluate three hormones that are associated with amenorrhea and infertility: follicle stimulating hormone, estradiol, and antimullerian hormone.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation to the Fistula Care Centre in Lilongwe for medical evaluation
2. Ability to consent for study participation in Chichewa
3. Female aged 18-45 years
4. Willingness to undergo pelvic ultrasound for assessment of pelvic organs

Exclusion Criteria:

1. No history of pregnancy
2. History of hysterectomy
3. Current pregnancy or pregnancy within the past six weeks
4. Seriously or terminally ill

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will be enrolling 100 Malawian women with obstetric fistula and 10 Malawian women without obstetric fistula.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cervical length | baseline

SECONDARY OUTCOMES:
Hormonal levels | baseline
  FSH, Estradiol, AMH

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wilkinson, MD, Study Director — University of North Carolina
Locations (1):
- Fistula Care Centre, Lilongwe, Malawi